CLINICAL TRIAL: NCT02595333
Title: Differences in Incision Pain and Uterine Contraction Pain After Cesarean Section Between Primary Section and Repeat Section
Brief Title: Incision Pain and Uterine Contraction Pain After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Obstetrics and Gynecology Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TT-Wang
Record Dates: First submitted 2015-10-26; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: C.Delivery; Surgery (Previous), Gynecological
Keywords: repeat cesarean section; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group SF1 (Experimental): primary cesarean section+postoperative analgesia with sufentanil plus flurbiprofen axetil group
  Interventions: Drug: Group SF1
- Group S1 (Experimental): primary cesarean section+postoperative analgesia with sufentanil group
  Interventions: Drug: Group S1
- Group SF2 (Experimental): repeated cesarean section+postoperative analgesia with sufentanil plus flurbiprofen axetil group
  Interventions: Drug: Group SF2
- Group S2 (Experimental): repeated cesarean section+postoperative analgesia with sufentanil group
  Interventions: Drug: Group S2

INTERVENTIONS:
Drug: Group SF1 — primary cesarean section+postoperative analgesia with sufentanil plus flurbiprofen axetil group
  Other Names: 1
  Arms: Group SF1
Drug: Group S1 — sufentanil was administered for analgesia in primary cesarean section
  Other Names: 2
  Arms: Group S1
Drug: Group SF2 — sufentanil and flurbiprofen was administered for analgesia in repeated cesarean section
  Other Names: 3
  Arms: Group SF2
Drug: Group S2 — sufentanil was administered for analgesia in repeated cesarean section
  Other Names: 4
  Arms: Group S2

SUMMARY:
This study aims to compare the pain degree between primary cesarean section and repeated cesarean section, and investigate the role of flurbiprofen axetil in postoperative analgesia, so as to provide reference for clinical practice.

DETAILED DESCRIPTION:
No premedication was given. The temperature of the operating room was maintained at 22˚ C. Patients were positioned supine with 15° left lateral tilt achieved using a wedge under the right buttock. Electrocardiograph(ECG), pulse oxygen saturation (SpO2), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and heart rate (HR) were monitored by one anesthesiologist (S/5 Anesthesia Monitor, GE Healthcare, Helsinki, Finland). Peripheral vein catheterization on the right hand was then performed, but no prehydration was given. A fixed volume of 500 ml hydroxyethyl starch solution was infused at the rate of 0.2 ml•kg-1•min-1, then Lactated Ringer's solution was infused at the same rate to the end of surgery. Combined spinal-epidural anesthesia was administered with patients in the left lateral position at the L3-4 vertebral interspace. A 16-gauge Tuohy needle was placed in the epidural space using loss of resistance to saline, then a 25-gauge Whitacre spinal needle was inserted through the Tuohy needle until the dura mater was punctured. Once free flow of clear cerebrospinal fluid (CSF) was observed in the spinal needle, 10 mg (2 mL) of isobaric bupivacaine 0.5% was diluted with CSF to 2.5 mL, then injected over 15-30 s. After placement and fixation of an epidural catheter, the patients were positioned supine with 15° left lateral tilt, and oxygen was given via nasal catheter at 2L.min-1. The sensory block level to cold was monitored every three minutes (1, 4, 7 and 10 min) with alcohol swabs and was recorded at the time point of 10 min. Hypotension was defined as SBP lower than 80% of the baseline value, and was treated with intravenous phenylephrine 100 µg as required. Intravenous atropine 0.3 mg was given for severe sinus bradycardia (HR < 50 beats/min). Surgery was allowed to start after the sensory block reached the T6 level; if this level was not achieved, patients were excluded from the study. For patients with inadequate sensory block, 1.5% lidocaine was given through the epidural catheter.

Four groups were divided based on surgical types and postoperative analgesia regimens, with 20 cases in each group: primary cesarean section + postoperative analgesia with sufentanil plus flurbiprofen axetil group(Group SF1), primary cesarean section+postoperative analgesia with sufentanil group (Group S1), repeated cesarean Section + postoperative analgesia with sufentanil plus flurbiprofen axetil group(Group SF2), and repeated cesarean section+ postoperative analgesia with sufentanil group(Group S2). Analgesia regimen: PCIA,100 ml; sufentanil 100 ug, ramosetron 0.3 mg, flurbiprofen axetil 100 mg (varied in groups); backgroup dosage 2 ml/h, PCA 2 ml each time, lock time 20 min. The scores of incision pain and uterine contraction pain 24 h, 48 h and 72 h after operation and the dose and pumping times of analgesia pump 24 h after operation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Eighty women undergoing elective cesarean section under general anesthesia were enrolled in this prospective observational study.

Exclusion Criteria:

* Diabetes controlled by insulin
* Preeclampsia
* Heart diseases
* History of taking drugs potentially affecting cardiovascular system.
* Patients fasted for at least 8 hours before surgery and no premedication was given

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The scores of incision pain and uterine contraction pain 24 h, 48 h and 72 h after operation | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, Study Director — Department of Anesthesiology, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China